CLINICAL TRIAL: NCT00547287
Title: Switching From Sildenafil Citrate to Tadalafil in Treatment of Erectile Dysfunction: Multinational Assessment of Treatment Preference
Brief Title: Studying the Preference of Tadalafil to Sildenafil in Men With Problems Getting an Erection Across Nations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ICOS Corporation (Industry)
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 7925; H6D-VI-LVFH
Record Dates: First submitted 2007-10-18; First posted 2007-10-22 (Estimated); Last update posted 2007-10-22 (Estimated); Status verified 2007-10

CONDITIONS: Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil; Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Currently prescribed dosage of sildenafil is continued until wash-out period.
  Interventions: Drug: sildenafil
- 2 (Active Comparator): 20 mg tadalafil given after one week sildenafil wash-out period.
  Interventions: Drug: tadalafil

INTERVENTIONS:
Drug: tadalafil — 20 mg tadalafil as needed by mouth no more than once a day for a 4 week initiation period and a 4 weeks treatment period.
  Other Names: LY450190; Cialis; IC351
  Arms: 2
Drug: sildenafil — Current dosage of sildenafil is continued for 4 weeks (no more than once a day) of treatment assessment then the wash-out period will begin.
  Arms: 1

SUMMARY:
Study to determine if men from around the world prefer sildenafil to tadalafil.

ELIGIBILITY:
Inclusion Criteria:

* Must be of legal age according to your country.
* Must have had a history of erectile dysfunction for at least 3 months.
* Must currently and have been using sildenafil for the last six weeks.
* Agree to not use any other ED treatment during the study.
* Anticipate the same female sexual partner for the study.

Exclusion Criteria:

* History of other primary sexual disorder
* Treatment with nitrates
* Have a penile implant or clinically significant penile deformity
* History of certain heart problems
* Do not meet certain lab value reference ranges

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2760 (Actual)
Dates: Start 2002-11; Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Patient choice of treatment (either sildenafil or tadalafil) for use in the extension phase | 14 weeks

SECONDARY OUTCOMES:
Assessment of sexual encounter attributes measured by the PAIRS scale including the Sexual Self-Confidence, Romance, and Time Pressure domains. | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo, Brazil

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com